CLINICAL TRIAL: NCT05291962
Title: Procedural Sedation for Pediatric Patients With Spinal Muscular Atrophy Undergoing Intrathecal Treatment
Brief Title: Procedural Sedation for Pediatric Patients With Spinal Muscular Atrophy
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Feyza Sever, Principal investigator, Ankara City Hospital Bilkent
Other Study IDs: 2019-159
Record Dates: First submitted 2022-02-08; First posted 2022-03-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Muscular Atrophy, Spinal; Child, Only; Anesthesia
Keywords: Spinal muscular atrophy; Procedural sedation; Children; Intratechal treatment
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Retrospective observational study — Data from anesthesia charts and electronic medical records of 14 patients with SMA type I, II and III who underwent procedural sedation,such as; the demographics data of the patients (age, gender, weight, American Society of Anesthesiologist (ASA) Physical Status), which anesthetic agent was used and their doeses, during of anesthesia, presence of scoliosis, by whom the procedure was performed etc. was reviewed.

SUMMARY:
Background and Aim: Spinal muscular atrophy (SMA) is a neuromuscular disease characterized by progressive symmetrical weakness and atrophy of proximal muscles causing from degeneration of anterior horn cells of spinal cord. Nusinersen must be administered intrathecally and this treatment is specially for spinal muscular atrophy. Procedural sedation is commonly enough for intrathecal treatment in children. In this retrospective study, the investigators aimed to present our experience in procedural sedation for the intrathecal treatment of patients with SMA 1,2 and 3 in our hospital.

DETAILED DESCRIPTION:
Design: This research is a retrospective obsevational study. Methods: After approval Institutional Review Board, data from anesthesia charts and electronic medical records of 14 patients with SMA type I, II and III who underwent procedural sedation,such as; the demographics data of the patients (age, gender, weight, American Society of Anesthesiologist (ASA) Physical Status), which anesthetic agent was used and their doeses, during of anesthesia, presence of scoliosis, by whom the procedure was performed etc. was reviewed. All our patients with SMA type II and III who underwent intrathecal treatment are given sedation with different combination of anesthetic agent. Due to peripheral intravenous line was placed previously, intravenous induction was performed in all of our patients For procedural sedation, anesthesiologists used different combination of midazolam, ketamine, propofol, fentanyl or remifentanyl, depending on the patient's requirement. They were oxygenated with a face mask or nasal cannula while their spontaneous breathing continues. All patients were recovered in the recovery room.

Statistical analysis: The data were analyzed by using SPSS Statistics Software (SPSS 24, Chicago, IL, USA) Descriptive statistics were used in this study. Mean and standart deviation were calculated for Age (year), Weight (kilogram), Midazolam Dose (mg/kg), Fentanyl Dose (mcg/kg), Remifentanyl Dose (mcg/kg), Propofol Dose (mg/kg), Ketamine Dose (mg/kg) and Length of Stay in Recovery Room (minute) and frequency analysis were made for the number of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients younger than 18 years old with SMA 1,2 and 3 who were to undergo intrathecal Nusinersen treatment were included in this study.

Exclusion Criteria:

* Patients whose procedures were performed under fluoroscopic guidance in the radiology unit were excluded from the study because their procedures were performed in another hospital.
* Patients without a diagnosis of SMA

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatric patients younger than 18 years old with SMA 1,2 and 3 who were to undergo intrathecal treatment under procedural sedation in our clinic
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Procedural sedation | 4 years (The data of the patients were retrospectively analyzed between July 2017 and December 2021.)
  The number of pediatric patients with SMA I,II and III who underwent intrathecal treatment required procedural sedation
Anesthetics use | 4 years (The data of the patients were retrospectively analyzed between July 2017 and December 2021.)
  The anesthetic agents and their doses that used during procedure
Age | 4 years (The data of the patients were retrospectively analyzed between July 2017 and December 2021.)
  Age in year
Gender | 4 years (The data of the patients were retrospectively analyzed between July 2017 and December 2021.)
  Gender as female/male
Weight | 4 years (The data of the patients were retrospectively analyzed between July 2017 and December 2021.)
  Weight in kilograms
American Society of Anesthesiologists (ASA) physical status | 4 years (The data of the patients were retrospectively analyzed between July 2017 and December 2021.)
  ASA score
Type of SMA | 4 years (The data of the patients were retrospectively analyzed between July 2017 and December 2021.)
  SMA I, SMA II and SMA III

SECONDARY OUTCOMES:
Presence of scoliosis | 4 years The data of the patients were retrospectively analyzed between July 2017 and December 2021.)(
  Yes or no
How many times intrathecal treatment was performed for each patient | 4 years The data of the patients were retrospectively analyzed between July 2017 and December 2021.)
  The number of intrathecal treatments was administered for each patient over 4 years was recorded.
By whom the procedure was performed | 4 years The data of the patients were retrospectively analyzed between July 2017 and December 2021.)
  It was recorded who performed the lumbar puncture procedure from a neurologist, neurosurgeon, or anesthesiologist.
Length of time spent in recovery room | 4 years The data of the patients were retrospectively analyzed between July 2017 and December 2021.)
  Recovery time in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Feyza Sever, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Feyza Sever, Ankara, Çankaya, Turkey (Türkiye)